CLINICAL TRIAL: NCT07133633
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tulisokibart in Participants With Radiographic Axial Spondyloarthritis (Ankylosing Spondylitis)
Brief Title: A Clinical Study of Tulisokibart (MK-7240) to Treat Radiographic Axial Spondyloarthritis (MK-7240-013)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7240-013; 2025-521059-21-00 (Registry Identifier: EU CT); U1111-1318-5807 (Registry Identifier: UTN); MK-7240-013 (Other: MSD)
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Radiographic Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- High-dose tulisokibart (Experimental): Participants receive a high dose of tulisokibart.
  Interventions: Drug: Tulisokibart
- Medium-dose tulisokibart (Experimental): Participants receive a medium dose of tulisokibart.
  Interventions: Drug: Tulisokibart
- Low-dose tulisokibart (Experimental): Participants receive a low dose of tulisokibart and are rerandomized at week 16 to a medium or high dose of tulisokibart.
  Interventions: Drug: Tulisokibart
- Placebo (Placebo Comparator): Participants receive a matched placebo dose and are rerandomized at week 16 to a medium or high dose of tulisokibart.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tulisokibart — Subcutaneous (SC) administration
  Other Names: MK-7240; PRA023
  Arms: High-dose tulisokibart; Low-dose tulisokibart; Medium-dose tulisokibart
Drug: Placebo — SC administration
  Arms: Placebo

SUMMARY:
Researchers are looking for new ways to treat radiographic axial spondyloarthritis (r-axSpA). R-axSpA is a type of arthritis that causes pain, stiffness, and inflammation (swelling) in the spine and joints in the pelvis (hip bone). Radiographic means the damage it causes can be seen on X-rays.

This study will help find out if a study medicine called tulisokibart can treat symptoms of r-axSpA. Researchers will look at different doses of tulisokibart.

Researchers want to know if at least one of the study doses of tulisokibart works better than a placebo to improve r-axSpA symptoms. A placebo looks like the study medicine but has no study medicine in it. Using a placebo helps researchers better understand the effects of the study medicine.

DETAILED DESCRIPTION:
This study consists of a 16-week Placebo-controlled Period and a 124-week Long-term Extension (LTE), which is composed of a 40-week Main Extension and an 84-week Optional Extension.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a clinical diagnosis of axial spondyloarthritis (axSpA) and meets the Assessment of SpondyloArthritis international Society (ASAS) classification criteria for axSpA including ≥3 months of back pain with age at symptom onset <45 years
* Meets the radiographic criterion of the modified New York criteria for ankylosing spondylitis (AS) as determined by central reading at Screening
* Has active disease at Screening and Randomization
* Has a history of inadequate response (IR)/intolerance to nonsteroidal anti-inflammatory drugs (NSAIDs) and is biologic disease-modifying antirheumatic drug (bDMARD)-naive, or has a history of IR/intolerance to up to a maximum of 2 bDMARD classes

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has any arthritis with onset before age 17 years or current diagnosis of inflammatory joint disease other than radiographic axial spondyloarthritis (r-axSpA) (such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis (PsA), systemic sclerosis, myositis, etc.), or any other conditions that may, in the judgment of the investigator, interfere with the assessment of r-axSpA
* Has a history of cancer (except fully treated non-melanoma skin cancers or cervical carcinoma in situ after complete surgical removal) within the last 5 years
* Has any active infection
* Has known allergies, hypersensitivity, or intolerance to tulisokibart or its excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2030-02-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Assessment of Spondyloarthritis International Society (ASAS) 40 Response at Week 16 | Week 16
  ASAS 40 is defined as a relative improvement of ≥40% and an absolute improvement of ≥2 units from baseline in ≥3 of 4 domains, with no deterioration in the fourth domain. The 4 domains include Patient Global Assessment (PtGA), total spinal pain, physical function, and morning stiffness. Each domain is measured on a 10-point numeric scale from 0 = no disease symptoms/impact to 10 = extreme disease symptoms/impact, with a higher score indicating more severe impairment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Ankylosing Spondylitis Disease Activity Score (ASDAS) <2.1 at Week 16 | Week 16
  ASDAS is a disease activity measure calculated from the assessments of total spinal pain, duration of morning stiffness, peripheral pain/swelling, PtGA, and high sensitivity C-reactive protein (hsCRP) as follows: 0.121 × total spinal pain (Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] question 2) + 0.110 × PtGA + 0.073 × peripheral pain/swelling (BASDAI question 3) + 0.058 × duration of morning stiffness (BASDAI question 6) + 0.579 × natural logarithm (ln) of (hsCRP + 1). ASDAS <2.1 indicates low disease activity and a higher score indicates greater disease activity.
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 16 | Baseline and Week 16
  The BASFI is a validated 10-item measure assessing individual-reported function (8 items) and ability to cope with everyday life (2 items) over the past week. Responses are recorded for each item on an 11-point numeric rating scale (NRS) from 0 "easy" to 10 "impossible". A mean score of the 10 items will be calculated to reflect the overall functional impairment, with higher scores indicating greater disability.
Change From Baseline in the Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Score for Spine at Week 16 | Baseline and Week 16
  The SPARCC MRI score for spine is a validated scoring system developed to assess inflammation in the spine related to axSpA. The 6 most abnormal discovertebral units are selected, and 3 consecutive sagittal slices are assessed. Each discovertebral unit is divided into 4 quadrants, scored as 1 if increased signal is present or 0 if normal, with a maximum of 12 points per discovertebral unit. Additional points are added for lesions that exhibit intense signal or deep (≥1 cm), increasing the maximum score per unit to 18. Summed over 6 slices, the maximum total score is 108. Higher scores indicate more extensive and/or intense spinal inflammation.
Change From Baseline in the SPARCC MRI Score for Sacroiliac Joint (SIJ) at Week 16 | Baseline and Week 16
  The SPARCC MRI score for SIJ is a validated scoring system to assess SIJ inflammation in axSpA. Six consecutive SIJ coronal slice images are assessed by dividing into 4 quadrants and scored as 1 if increased signal is present or 0 if normal, with a maximum of 8 points per slice for both joints. Additional points are added for lesions that exhibit intense signal or deep (≥1 cm), increasing the maximum score per unit to 12. Summed over 6 slices, the maximum total score is 72. Higher scores indicate more extensive and/or intense SIJ inflammation.
Change From Baseline in Total Spinal Pain Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Question 2 at Week 16 | Baseline and Week 16
  The BASDAI is a validated 6-item questionnaire used to assess disease activity in radiographic axial spondyloarthritis. It assesses individual-reported fatigue, total spinal pain, peripheral pain/swelling, tenderness, intensity of morning stiffness, and duration of morning stiffness over the past week. To access individual-reported total spinal pain experienced over the past week, participants are asked BADSAI question 2, "How would you describe the overall level of ankylosing spondylitis neck, back, or hip pain you have had?" Responses are recorded on an 11-point NRS ranging from 0 "none" to 10 "very severe." Higher score indicates more severe total spinal pain.
Change From Baseline in Nocturnal Spinal Pain at Week 16 | Baseline and Week 16
  The NRS is an 11-point scale (numeric version of the visual analog scale) to assess the pain intensity in individuals who can self-report. Participants will be asked to report their average nighttime spinal pain over the past week on an 11-point NRS. The score range is from 0 "no pain" to 10 "most severe pain." Higher score indicates more severe nocturnal spinal pain.
Change From Baseline in Assessment of Spondyloarthritis International Society Health Index (ASAS HI) at Week 16 | Baseline and Week 16
  The ASAS HI assesses overall functioning and health and is a validated 17-item individual-reported measure of pain, emotional functions, sleep, sexual function, mobility, self-care, and community life, with response options of "I agree" (1) or "I do not agree" (0). The ASAS HI is a total summary score ranging from 0 to 17 with a lower score indicating a better and a higher score indicating an inferior health status.
Change From Baseline in Short Form-36 Health Survey (SF-36) Physical Component Summary (PCS) at Week 16 | Baseline and Week 16
  The SF-36 is a widely used general health status questionnaire that assesses 8 domains of functional health and well-being: physical functioning, role limitations due to physical health problems, bodily pain, social functioning, mental health, role limitations due to emotional problems, vitality, and general health perceptions. The PCS score is a composite score derived from the SF-36 that summarizes the physical health aspects of the survey. It combines information primarily from the physical domains (physical functioning, role limitations due to physical health problems, bodily pain, and general health perceptions). All SF-36 scores range from 0 = worst health state to 100 = best health state, with higher scores indicating a better health-related quality of life (QoL).
Change From Baseline in BASDAI at Week 16 | Baseline and Week 16
  The BASDAI is a validated 6-item measure, assessing individual-reported fatigue, total spinal pain, peripheral pain/swelling, tenderness, intensity of morning stiffness, and duration of morning stiffness over the past week. Responses are recorded for each item on an 11-point NRS from 0 "none" to 10 "very severe." BASDAI is calculated by averaging the response for question 5 and question 6, adding this result to the sum of question 1 through question 4, and then dividing the result by 5. A higher score indicates greater disease activity.
Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 16 in the Subgroup of Participants With Enthesitis (MASES>0) at Baseline | Baseline and Week 16
  The MASES is a validated method to assess peripheral enthesitis in axSpA. It assesses pain on palpation at the following anatomic sites: first costochondral joint (right & left); seventh costochondral joint (right & left); anterior superior iliac spine (right & left); iliac crest (right & left); posterior superior iliac spine (right & left); fifth lumbar spinous process; Achilles tendon, proximal insertion (right & left). Each site is scored based on participant response as either 0 (nontender) or 1 (tender), the final score ranges from 0 (absence of enthesitis) up to a score of 13 (enthesitis present at all sites). Injected enthesitis sites will be considered not assessable for 90 days from the time of the injection. Higher score indicates more tender or inflamed enthesitis sites. Resolution of enthesitis is defined as MASES score equal to zero.
Change From Baseline in Bath Ankylosing Spondylitis Metrology Index Linear (BASMI lin) at Week 16 | Baseline and Week 16
  The BASMI lin is a validated tool to assess mobility in axSpA. The BASMI lin evaluates the range in centimeters of 5 components of hip and spinal mobility (components: tragus-to-wall, lateral lumbar flexion, cervical rotation angle, lumbar flexion, and maximal intermalleolar distance). For tragus to wall, lateral lumber flexion, and cervical rotation angle, the average measurements from left and right would be used as the component score. Component score range is from 0 (no mobility limitation) to 10 (very severe mobility limitation). Higher score indicates more severe mobility limitation.
Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) at Week 16 | Baseline and Week 16
  The FACIT-Fatigue is a validated 13-item measure that assesses individual-reported fatigue and its impact on daily activities and function during usual activities over the past week. Responses are recorded on a 5-point Likert scale (0 = not at all to 4 = very much), individual item scores are then summed to provide the final score with range from 0 (worst score/extreme fatigue) to 52 (best score/no or minimal fatigue). Higher total scores represent lower levels of fatigue.
Number of Participants With One or More Adverse Events (AEs) | Up to approximately 154 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 140 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (73):
- United States (28):
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Chandler ( Site 0036), Chandler, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Flagstaff ( Site 0021), Flagstaff, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C. - Gilbert ( Site 0022), Gilbert, Arizona
  - AARA Arizona Arthritis & Rheumatology Associates, P.C. - Glendale ( Site 0056), Glendale, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C. - Tucson ( Site 0025), Tucson, Arizona
  - TriWest Research Associates - Chula Vista ( Site 0013), Chula Vista, California
  - Newport Huntington Medical Group ( Site 0005), Huntington Beach, California
  - Cohen Medical Centers ( Site 0034), Thousand Oaks, California
  - Inland Rheumatology Clinical Trials, Inc. ( Site 0002), Upland, California
  - Arthritis and Rheumatic Disease Specialties ( Site 0016), Aventura, Florida
  - GNP Research - Hollywood ( Site 0020), Cooper City, Florida
  - Innovation Medical Research Center ( Site 0012), Palmetto Bay, Florida
  - Chicago Arthritis & Regenerative Medicine ( Site 0042), Chicago, Illinois
  - Willow Rheumatology and Wellness, PLLC ( Site 0035), Willowbrook, Illinois
  - Arthritis and Rheumatism Associates - Rockville ( Site 0019), Rockville, Maryland
  - Kansas City Physician Partners ( Site 0027), Kansas City, Missouri
  - Velocity Clinical Research - West County Rheumatology, St. Louis ( Site 0038), St Louis, Missouri
  - Physician Research Collaboration, LLC ( Site 0057), Lincoln, Nebraska
  - Inspire Santa Fe Medical Group ( Site 0011), Santa Fe, New Mexico
  - Altoona Center for Clinical Research ( Site 0004), Duncansville, Pennsylvania
  - Perelman Center for Advanced Medicine ( Site 0060), Philadelphia, Pennsylvania
  - AARA Clinical Research - Murfreesboro Medical Clinic ( Site 0029), Murfreesboro, Tennessee
  - Arthritis Care of Texas ( Site 0048), Corpus Christi, Texas
  - Lone Star Arthritis & Rheumatology Associates, P.C. ( Site 0028), Fort Worth, Texas
  - Provecta Research Network LLC ( Site 0054), Houston, Texas
  - AARA Clinical Research - Lone Star Arthritis and Rheumatology Associates - Irving ( Site 0032), Irving, Texas
  - Epic Medical Research ( Site 0061), Red Oak, Texas
  - DM Clinical Research - TRA ( Site 0010), Tomball, Texas
- CMIP-CENTRO MINEIRO DE PESQUISA ( Site 1999), Juiz de Fora, Minas Gerais, Brazil
- Canada (2):
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc. ( Site 0200), Québec, Quebec
  - Centre de Recherche Musculo-Squelettique ( Site 0202), Trois-Rivières, Quebec
- China (9):
  - The First Afflilated Hospital of Bengbu Medical College ( Site 3119), Bengbu, Anhui
  - Chinese Academy of Medical Science Peking Union Medical College Hospital ( Site 3100), Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital ( Site 3110), Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-Sen University ( Site 3114), Guangzhou, Guangdong
  - The First Affiliated Hospital of Henan University of Science &Technology ( Site 3121), Luoyang, Henan
  - Pingxiang People's Hospital ( Site 3115), Pingxiang, Jiangxi
  - The First Hospital Of Jilin University ( Site 3103), Changchun, Jilin
  - PEOPLE'S HOSPITAL OF XINJIANG UYGUR AUTONOMOUS REGION ( Site 3124), Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University ( Site 3123), Kunming, Yunnan
- Colombia (3):
  - Clinica de la Costa S.A.S. ( Site 2202), Barranquilla, Atlántico
  - CIREEM SAS ( Site 2204), Bogota, Cundinamarca
  - Fundación Valle del Lili ( Site 2201), Cali, Valle del Cauca Department
- Germany (3):
  - Medicover München Ost MVZ ( Site 0611), Munich, Bavaria
  - Rheumatologische Schwerpunktpraxis ( Site 0605), Berlin
  - HRF II - Hamburger Rheuma Forschungszentrum II MVZ für Rheumatologie und Autoimmunmedizin Hamburg G ( Site 0604), Hamburg
- Netherlands (2):
  - Zuyderland Medical Centre ( Site 1100), Heerlen, Limburg
  - Amsterdam UMC ( Site 1101), Amsterdam, North Holland
- Poland (5):
  - MICS Centrum Medyczne Bydgoszcz ( Site 1206), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr 2 im. dr J. Biziela w Bydgoszczy ( Site 1203), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun ( Site 1202), Torun, Kuyavian-Pomeranian Voivodeship
  - Zespół Poradni Specjalistycznych Reumed Filia nr 1 Wallenroda ( Site 1201), Lublin, Lublin Voivodeship
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im.Prof. El. Reicher-ul.Spartanska 1 ( Site 1205), Warsaw, Masovian Voivodeship
- South Korea (2):
  - Hanyang University Seoul Hospital ( Site 2800), Seoul
  - Kyung Hee University Hosptial at Gangdong ( Site 2802), Seoul
- Taiwan (6):
  - Taipei Medical University Shuang Ho Hospital ( Site 2900), New Taipei City, New Taipei
  - Kaohsiung Veterans General Hospital ( Site 2905), Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 2908), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 2903), Tainan
  - Taipei Veterans General Hospital ( Site 2906), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 2904), Taoyuan District
- Ukraine (9):
  - Communal Nonprofit Enterprise Cherkasy Regional Hospital of Cherkasy Oblast Council ( Site 1704), Cherkasy, Chernivetska Oblast
  - Municipal Public Non-Profit Enterprise "City Clinical Hospital №1 of the Ivano-Frankivsk City Counc ( Site 1705), Ukraine, Ivano-Frankivsk Oblast
  - Municipal Non-Profit Enterprise "Khmelnytskyi Regional Hospital" of Khmelnytskyi Regional Council ( Site 1713), Khmelnytskiy, Khmelnytskyi Oblast
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical" ( Site 1715), Kyiv, Kyivska Oblast
  - Lviv Clin Hospital of Planned Treatment Rehabilitation Palliative Care ( Site 1710), Lviv, Lviv Oblast
  - ME "Ternopil Regional Clinical Hospital of Ternopil Regional Council" ( Site 1707), Ternopil, Ternopil Oblast
  - Municipal Nonprofit Enterprise "Vinnytsia Regional Clinical Hospital n.a. M. I. Pyrohov of Vinnytsia ( Site 1700), Vinnytsa, Vinnytsia Oblast
  - Kyiv Railway Clinical Hospital No.2 of Branch Health Center of the Public Joint Stock Company Ukrain ( Site 1701), Kyiv
  - Medical Center "Universal Clinic "Oberig" of Limited Liability Company "Kapytal" ( Site 1706), Kyiv
- United Kingdom (3):
  - Norfolk & Norwich University Hospital NHS Foundation Trust ( Site 1800), Norwich, Norfolk
  - Royal United Hospital Bath NHS Foundation Trust ( Site 1803), Bath, Somerset
  - Barnet Hospital ( Site 1806), Barnet

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com